CLINICAL TRIAL: NCT03027921
Title: Validation in a Non-targeted Population (Screening) of Single Ultrasound Doppler Signs of Liver Fibrosis
Brief Title: Validation in a Non-targeted Population of Single Ultrasound Doppler Signs of Liver Fibrosis
Acronym: DECHO2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 49RC16_0164
Record Dates: First submitted 2017-01-19; First posted 2017-01-23 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2017-01

CONDITIONS: Cirrhosis
MeSH Terms: conditions — Fibrosis

ARMS (1):
- hepatic ultrasound (Experimental): all patients will have hepatic ultrasound
  Interventions: Other: elastography

INTERVENTIONS:
Other: elastography

SUMMARY:
The diagnosis of liver fibrosis lesions remains an important issue in patients with chronic liver diseases. The early detection of fibrosis is important for determining disease progression and postponing the evolution of chronic hepatitis into cirrhosis via the implementation of prompt and specific treatment. However, as chronic liver disease can remain asymptomatic for a long time, numerous cirrhotic patients are diagnosed belatedly, when life-threatening complications start appearing.

Noninvasive methods for liver fibrosis diagnosis have been developed over the last decade. In this setting, blood fibrosis tests and transient elastography have been shown to be accurate, and are now commonly used as first-intention tests for liver fibrosis diagnosis in chronic liver diseases. However, these tests are usually performed by a hepatologist to whom the patient has been referred following the appearance of symptoms suggestive of chronic liver disease. Thus the number of patient diagnosed early by these new tools, that is in the period before symptoms start appearing and during which preventative measures may be particularly beneficial, remains quite low in relation to the prevalence of the disease. This prevalence has been estimated to 0.5 to 2.8 % in general population.

Many studies have identified the value of hemodynamic and morphological ultrasound parameter in providing information on liver fibrosis degree. Moreover, abdominal ultrasound is widely used for various symptoms, and thus could be an excellent way to detect patients with signs evoking liver fibrosis or cirrhosis, who could then be referred to a liver specialist for confirmation of the diagnosis by blood fibrosis tests and/or transient elastography. To be feasible during a nonspecific US examination, and by any radiologist, these signs should be easy and quick to collect. Addition of a quick measure of hepatic stiffness could increase the screening interest of ultrasound examination.

The main aim of the present study was thus to validate 3 simple US signs in patients referred for ultrasound abdominal examination for reasons other than suspicion of liver disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred to an ultrasound unit for abdominal US examination, whatever the indication.
* Patient with Social Security

Exclusion Criteria:

* Age <18 years
* Previously identified chronic liver disease
* Hematological disease
* Patient under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2017-02; Primary Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Evaluate the number of patients with severe hepatic fibrosis detected by a progressive algorithm combining simple ultrasound signs of fibrosis and measurement of liver hardness in a non-suspect population of chronic hepatopathies. | 6 month

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Angers, Angers, France, France